CLINICAL TRIAL: NCT04997369
Title: Feasibility and Multicenter Assessment of Catheter-less Water Vapor Therapy (Rezum) for the Treatment of Benign Prostatic Hyperplasia (BPH)
Brief Title: Catheterless Water Vapor Therapy for the Treatment of BPH
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator changing locations.
Sponsor: Northwell Health (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20-02021474
Record Dates: First submitted 2021-07-29; First posted 2021-08-09 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Water Vapor Therapy
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Catheterless group (Experimental)
  Interventions: Device: Rezum

INTERVENTIONS:
Device: Rezum — The Rezum system is an ablative procedure for patients with benign prostatic hyperplasia (BPH).
  Other Names: Water vapor therapy

SUMMARY:
The Rezum system is an ablative procedure for patients with benign prostatic hyperplasia (BPH). One of the limitations of the technology is the need for post-operative catheterization up to 5 days. The aim of this study is to assess the feasibility of employing Catheterless Rezum post-operatively in patients with normal or strong bladder contractility. Upon a positive outcome of interim analysis, the effectiveness of Catheterless Rezum will be assessed at five sites for the multicenter phase.

ELIGIBILITY:
Inclusion Criteria:

* Male subject of 40 - 80 years of age
* Has provided informed consent
* Has a diagnosis of bladder outlet obstruction due to benign prostatic enlargement
* Able to complete self-administered questionnaires
* Is a surgical candidate for Rezum
* Has medical record documentation of Qmax < 15 ml/s
* Has medical record documentation of prostate volume from 30-80 ml by transrectal ultrasound (TRUS)
* Has a bladder contractility index score ≥ 100, calculated by detrusor pressure at Qmax (pDet@qmax) + (5xQmax).
* Willing to undergo pressure-flow studies to calculate BCI prior to surgical intervention.
* Has serum creatinine within the normal range.
* Able to perform intermittent catheterization.

Exclusion Criteria:

* Has a life expectancy < 2 years
* Is currently enrolled in or plans to enroll in any concurrent drug or device study
* Has an active infection (e.g., urinary tract infection or prostatitis)
* Has a diagnosis of or has received treatment for chronic prostatitis or chronic pelvic pain syndrome (e.g., nonbacterial chronic prostatitis)
* Has been diagnosed with a urethral stricture or bladder neck contracture within the last 180 days
* Has been diagnosed with 2 or more urethral strictures and/or bladder neck contractures within 5 years
* Has a diagnosis of lichen sclerosis
* Has a diagnosis of neurogenic bladder or other neurologic disorder that affects bladder function
* Has a diagnosis of polyneuropathy (e.g., diabetic)
* Has a history of lower urinary tract surgery
* Has a diagnosis of stress urinary incontinence that requires treatment or daily pad or device use
* Has an inability to perform intermittent self-catheterization
* Has been catheterized or has a post-void residual (PVR) of > 400 ml in the 14 days prior to the surgical procedure
* Has a current diagnosis of bladder stones

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Catheterless Rezum as measured by changes in the International Prostate Symptom Score (IPSS). | Baseline, 36 months
  The outcome will be assessed based on a 6.0-point average improvement in the IPSS score. Higher scores indicate greater symptom severity and lower scores indicate less symptom severity.
Feasibility of Catheterless Rezum as measured by changes in the maximum urinary flow rate (Qmax). | Baseline, 36 months
  The outcome will be assessed based on a 2.5-point average improvement in Qmax compared to baseline. Higher Qmax values indicate less urinary obstruction while lower Qmax values correspond to increased urinary obstruction.

SECONDARY OUTCOMES:
Changes in urinary symptoms as measured by changes in IPSS. | Baseline, 36 months
  The outcome will be assessed based on a 6.0-point average improvement in the IPSS score. Higher scores indicate greater symptom severity and lower scores indicate less symptom severity.
Changes in urinary symptoms as measured by changes in Qmax at 36 months | Baseline, 36 months
  The outcome will be assessed based on a 2.5-point average improvement in Qmax compared to baseline. Higher Qmax values indicate less urinary obstruction while lower Qmax values correspond to increased urinary obstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Chughtai, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No